CLINICAL TRIAL: NCT05698784
Title: Relevance of 123 I-FP-CIT SPECT Prescriptions for the Diagnosis of Parkinsonian Syndromes
Brief Title: 123 I-FP-CIT SPECT Prescriptions for Parkinsonian Syndromes
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Centre Hospitalier Universitaire de la Guadeloupe (Other)
Responsible Party: Sponsor
Other Study IDs: CLEA-2019-75
Record Dates: First submitted 2023-01-16; First posted 2023-01-26 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-01

CONDITIONS: Parkinson

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group a "inappropriate": In the "inappropriate" , we placed prescriptions with no indication, 123I-FP-CIT SPECT
- Group b "uncertain": In the "uncertain", we did not have sufficient data to determine with certainty whether this was an inappropriate or relevant indication.
- Group c "relevant": In the "relevant" , the prescriptions concerned the differential diagnosis between neurodegenerative parkinsonism and secondary parkinsonian syndromes

SUMMARY:
123I-FP-CIT SPECT (DaTSCAN®) allows to detect presynaptic dopamine neuronal denervation. It is recommended to differentiate neurodegenerative parkinsonism from secondary parkinsonian syndromes or from essential tremor, and to distinguish patients with suspected dementia with Lewy bodies and those with other subtypes of dementia. The aim of this retrospective study was to evaluate the relevance of 123I-FP-CIT SPECT prescriptions, the profile of prescribers and the evolution of the prescription rate over a ten-year period.

DETAILED DESCRIPTION:
the investigators included 723 patients in this retrospective study between February 2009 and May 2019, in the nuclear medicine Department of Avicenne University Hospital. No patients were excluded. Demographic, clinical, brain imaging, and 123I-FP-CIT SPECT data were collected from medical records. The study was conducted in accordance with the Declaration of Helsinki, and approved by the Institutional Ethics Committee (CLEA-2019-75).

Regarding the relevance of the indications, the investigators have defined three groups: " inappropriate ", "uncertain " and " relevant ", also respectively named (a), (b) and (c) groups.

In the "inappropriate" group (a), the investigators placed prescriptions with no indication, 123I-FP-CIT SPECT requested to confirm a PS clinically evident, and those prescribed for isolated cognitive-behavioral disturbances with no PS or differential diagnosis mentioned.

In the "uncertain" group (b), the investigators did not have sufficient data to determine with certainty whether this was an inappropriate or relevant indication.

In the "relevant" group (c), the prescriptions concerned the differential diagnosis between neurodegenerative parkinsonism and secondary parkinsonian syndromes (for instance post-neuroleptics) or other doubtful disorders (Alzheimer's disease, essential tremor), clinically uncertain PS (such as an isolated asymmetric resting tremor without akinesia or lead-pipe rigidity) and PD of atypical evolution.

Data were presented as mean (standard deviation) for numeric variables and as count (percentage) for categorical variables. To compare demographic, clinical and paraclinical data, and the distribution of prescribers between the three groups (i.e. inappropriate (a), uncertain (b) and relevant (c)), one-factor analysis of variance (ANOVA) was used for numerical variables and Fisher's exact test for categorical variables. To identify which groups differed from each other, post hoc comparisons were made using the Tukey test for numeric variables and the Fisher pairwise exact test followed by the Benjamini-Hochberg correction to account for multiple testing, for categorical variables. For all tests, the significance level was set at p < 0.05. All data were analyzed using R software (version 3.6.1, R Core Team).

ELIGIBILITY:
Inclusion Criteria:

* Parkinsonian patients who benefited from a 123I-FP-CIT SPECT

Exclusion criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Parkinsonian patients who benefited from a 123I-FP-CIT SPECT ,
Sampling Method: Non-Probability Sample
Enrollment: 723 (Actual)
Dates: Start 2019-06 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Evaluate the relevance of 123I-FP-CIT SPECT prescriptions | February 2009 - May 2019
  Regarding the relevance of the indications, we have defined three groups: " inappropriate ", "uncertain " and " relevant ", also respectively named (a), (b) and (c) groups.
  To identify which groups differed from each other, post hoc comparisons were made using the Tukey test for numeric variables and the Fisher pairwise exact test followed by the Benjamini-Hochberg correction to account for multiple testing, for categorical variables. For all tests.

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand DEGOS, MD, PhD, Study Director — Hopital Avicenne
Locations (1):
- Hôpital Avicenne, Bobigny, France